CLINICAL TRIAL: NCT00914134
Title: Effect of Duodenal Levodopa Infusion on Quality of Life and Autonomic Dysfunction in Patients With Parkinson's Disease
Brief Title: Duodenal Levodopa Infusion, Quality of Life and Autonomic Nervous System in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Helsinki (Other)
Collaborators: Solvay Pharmaceuticals (Industry)
Responsible Party: Eero Pekkonen, Helsinki University Central Hospital, Department of Neurology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PDAUT2009
Record Dates: First submitted 2009-06-01; First posted 2009-06-04 (Estimated); Last update posted 2011-02-24 (Estimated); Status verified 2011-02

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Autonomic nervous system; Levodopa infusion
MeSH Terms: conditions — Parkinson Disease | interventions — carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Levodopa Infusion (Experimental): Patients with advanced Parkinson's disease and motor fluctuations that cannot be adequately controlled with oral medication.
  Interventions: Drug: Levodopa infusion

INTERVENTIONS:
Drug: Levodopa infusion — Naso-duodenal infusion line is inserted in fluoroscopy control. Levodopa infusion is then tested approximately 5 days. If patient responds favorably to the treatment, PEG-infusion line is inserted in gastroscopy control and patient is followed in hospital for 2 to 4 days to ensure stability of the infusion line. The dosage is individually adjusted, starting dose is estimated from earlier oral levodopa dose.
  Other Names: Duodopa

SUMMARY:
The aim of the study is to assess the effect of continuous levodopa infusion on autonomic nervous system in patients with Parkinson's Disease (PD), blood pressure regulation and sweating. The investigators' hypothesis is that levodopa infusion may alleviate hyperhidrosis and orthostatic hypotension.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is one of the most common neurodegenerative disorders with increasing prevalence because of aging population. The main symptoms include rigidity, hypokinesia, tremor and impaired balance, but the disease also causes autonomic dysfunction. Motor fluctuations are common treatment related problems in PD, around 50-70% of patients treated with levodopa finally develop motor fluctuations. Continuous duodenal levodopa infusion has been effective in the treatment of motor dysfunction in advanced PD. However, little is known of its effects on autonomic nervous system.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease: diagnosis made at least five years earlier
* Positive response to levodopa
* Motor fluctuations that cannot be adequately controlled with oral medication
* No signs or symptoms of cerebellar dysfunction or vascular parkinsonism

Exclusion Criteria:

* Severe cognitive symptoms
* Glaucoma
* Severe arrythmias
* Severe asthma or COPD
* Heart, liver or kidney failure
* No significant vascular lesions in brain MRI imaging.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-04; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
Orthostatic blood pressure change | Before levodopa infusion, after 3-5 days of levodopa infusion and 2 months after levodopa infusion was started

SECONDARY OUTCOMES:
Sweating measured by evaporimeter | Before levodopa infusion, after 3-5 days of levodopa infusion, 2 months after levodopa infusion was started
Autonomic nervous system symptoms questionnaire (NMSS) | Before levodopa infusion and 2 months after levodopa infusion was started
Quality of life questionnaire (PDQ-39) | Before levodopa infusion and 2 months after levodopa infusion was started

CONTACTS AND LOCATIONS:
Overall Officials: Eero Pekkonen, MD, PhD, Study Director — Helsinki University Central Hospital, Department of Neurology
Locations (1):
- Helsinki University Central Hospital, Department of Neurology, Helsinki, Finland